CLINICAL TRIAL: NCT04220684
Title: A Phase I Clinical Trial Testing the Safety of IL-21-Expanded, Off-the-shelf, Third-party Natural Killer Cells (KDS-1001) for the Induction of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Trial Testing Safety of IL-21 NK Cells for Induction of R/R AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumithira Vasu (Other)
Collaborators: Kiadis Pharma (Industry)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18336; NCI-2019-05150 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-09-26; First posted 2020-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Allogeneic Stem Cell Transplant Recipient; Blasts 10 Percent or More of Bone Marrow Nucleated Cells; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cytarabine; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conditioning Regimen (Experimental): Fludarabine 30 mg/m2/day (day -6 to day -2) and Cytarabine 2g/ m2/day (days -6 to day -2)
  Interventions: Drug: Cytarabine Hydrochloride; Drug: Fludarabine
- Induction (Experimental): Six doses of third-party-donor mbIL-21 expanded (KDS-1001) cells given thrice weekly for two weeks. Days may vary and KDS-1001 can be given from days 0 to 21
  Interventions: Biological: Membrane-bound Interleukin-21-Expanded Haploidentical Natural Killer Cells

INTERVENTIONS:
Drug: Cytarabine Hydrochloride — Given IV
  Other Names: Ara-C HCl; Arabinosylcytosine Hydrochloride; Aracytidine Hydrochloride; CHX-3311; Cytosar Hydrochloride; Cytosine Arabinosine Hydrochloride; U-19920A
  Arms: Conditioning Regimen
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Conditioning Regimen
Biological: Membrane-bound Interleukin-21-Expanded Haploidentical Natural Killer Cells — Given via infusion
  Other Names: (mbIL21)-expanded Haploidentical NK Cells; Donor mbIL21-expanded NK Cells; mbIL21-expanded Haploidentical NK Cells
  Arms: Induction

SUMMARY:
This phase I trial studies the side effects of donor natural killer (NK) cell therapy in treating patients with acute myeloid leukemia that has come back (recurrent) or has not responded to treatment (refractory). Natural killer cells are a type of immune cell. Immunotherapy with genetically modified NK cells from donors may induce changes in the body's immune system and may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of adoptive NK cell therapy using membrane-bound interleukin-21 (mbIL21)-expanded, off-the-shelf, third-party donor-derived NK cells in patients with relapsed/refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. Estimate the complete response (CR, CR with incomplete hematologic recovery [CRi] & morphologic leukemia-free state [MLFS]).

II. Estimate the median relapse free survival. III. Estimate the median time to neutrophil and platelet count recovery. IV. Estimate the median duration of remission. V. Estimate the incidence of infectious complications. VI. Estimate percentage of patients receiving this regimen who are rendered transplant-eligible.

CORRELATIVE OBJECTIVES:

I. Determine the persistence of ex-vivo expanded, off-the-shelf, third-party NK cells.

II. Characterize in vivo expansion of third-party NK cells and if it differs based on the conditioning regimen as defined by NK chimerism assay.

III. Determine the immunophenotype and function of expanded cells. IV. Chimerism analysis in patients who have had post-transplant relapses.

OUTLINE: This is a dose-escalation study of membrane-bound interleukin-21-expanded haploidentical natural killer cells.

INDUCTION: Patients receive fludarabine intravenously (IV) and cytarabine IV on days -6 to -2 in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients who are >= 60 years old, unable/unwilling to tolerate intensive chemotherapy, or disease insensitive to cytarabine (tp53, TET2 mutations) receive fludarabine IV on days -5 to -2 and decitabine IV on days -6 to -2 in the absence of disease progression or unacceptable toxicity.

All patients receive membrane-bound interleukin-21-expanded haploidentical natural killer cells via infusion on days 0, 2, 4, 7, 9, and 11.

After completion of study treatment, patients are followed up to day 56.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria for Induction Phase

* Primary Relapsed AML including
* Relapsed AML after allogeneic stem cells
* Isolated CNS or extramedullary disease (Note: a response monitoring plan must be developed a priori for subjects with extramedullary disease)
* 1-3 prior lines of therapy which includes chemotherapy, hypomethylating agents, venetoclax or targeted therapy.
* Patient weight ≥ 42 kg
* Performance status: Karnofsky or Lansky Performance Scale (PS) greater or equal to 70, or, ECOG score 0-2.
* Renal function: Serum creatinine ≤ 2 mg/dl and/or creatinine clearance greater or equal than 40 cc/min.
* Pulmonary function: FEV1, FVC and DLCO ≥ 50% of expected, corrected for hemoglobin.
* Liver function: Total bilirubin ≤ 2 mg/dl or ≤ 2.5 x ULN for age (unless Gilbert's syndrome) and SGPT (ALT) ≤ 2.5 x ULN for age.
* Cardiac function: left ventricular ejection fraction ≥ 40%.
* CNS: Patients with seizure disorder are eligible if seizures well controlled.
* Negative serum test to rule out pregnancy within 2 weeks prior to enrollment in females of childbearing potential (non-childbearing potential defined as premenarchal, greater than one year post-menopausal, or surgically sterilized).
* Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator.
* Ability to understand and willingness to sign the written informed consent document.
* Negative serology for human immunodeficiency virus (HIV).
* Patients on hydrocortisone for adrenal insufficiency or on inhaled or topical steroids are eligible.

Maintenance Phase: Patients that complete induction therapy and who achieve a CR/CRi/PR within the designated follow-up period and who are ineligible, unable or unwilling to undergo HSCT; these patients will not receive fludarabine or cytarabine.

Exclusion Criteria for Induction Phase:

* Investigational therapies in the 3 weeks prior to beginning treatment on this protocol.
* Patients receiving any concurrent therapy including but not limited to chemotherapy, targeted therapy, radiation therapy, or immunotherapy for R/R AML.
* Any comorbidities that in the opinion of the investigator will preclude receiving fludarabine or cytarabine.
* Uncontrolled infection, defined as an infection which has not resolved spontaneously or does not show evidence of significant resolution after initiating appropriate therapy. Asymptomatic viremia such as CMV, HPV, BK virus, HCV, HBV etc. is NOT considered as an exclusion criteria.
* Uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease.
* Active GVHD
* Prednisone dose is > 20 mg/day or >0.25mg/kg, whichever is higher will be excluded.
* Patients with donor-specific antibodies with MFI > 5000 will be ineligible
* Maintenance Phase: Patients must continue to meet exclusion criteria as defined in Section 4.4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of membrane-bound interleukin-21-expanded haploidentical natural killer (NK) cells | Up to 63 days
  The MTD will be defined as the highest safely tolerated dose where at most one patient in six experiences dose-limiting toxicity (DLT) during DLT observation period. DLT is defined as any steroid refractory acute graft versus host disease.
Incidence of adverse events | Up to day 28
  Toxicities will be assessed by type and grade using Common Terminology Criteria for Adverse Events version 5.0 and displayed in summary form by cohort and overall. Toxicities will be summarized and reported regardless of attribution and also only those attributed to NK cells.

SECONDARY OUTCOMES:
Complete response (CR) | Up to day 56
  Response rate with a 95% confidence interval (CI) will be reported for all evaluable patients, assuming a binomial distribution. Response rate will also be reported for those who received all 6 doses of NK cells.
CR with incomplete hematologic recovery | Up to day 56
  Response rate with a 95% CI will be reported for all evaluable patients, assuming a binomial distribution. Response rate will also be reported for those who received all 6 doses of NK cells.
Morphologic leukemia-free state | Up to day 56
  Response rate with a 95% CI will be reported for all evaluable patients, assuming a binomial distribution. Response rate will also be reported for those who received all 6 doses of NK cells.
Median relapse free survival | Up to day 56
  Will use descriptive statistics to summarize the demographic and clinical characteristics of the patients on this study.
Median time to neutrophil and platelet count recovery | Up to day 56
  Will use descriptive statistics to summarize the demographic and clinical characteristics of the patients on this study.
Median duration of remission | Up to day 56
  Will use descriptive statistics to summarize the demographic and clinical characteristics of the patients on this study.
Incidence of infectious complications | Up to day 56
  Will use descriptive statistics to summarize the demographic and clinical characteristics of the patients on this study.
Percentage of patients receiving the regimen who are rendered transplant-eligible | Up to day 56
  Will use descriptive statistics to summarize the demographic and clinical characteristics of the patients on this study.

OTHER OUTCOMES:
Identification of In-vivo expansion of NK cells | Up to day 56
  Peripheral blood will be obtained before therapy, during the NK cell treatment period, and after NK cell treatment. The studies may include flow cytometry analyses and sorting and molecular studies. Donor NK-cell expansion will be defined as an absolute circulating donor-derived NK cell count that increases above the post-infusion level.
Chimerism analysis to determine origin and number of circulating NK cells | Up to day 56
  Chimerism may be determined by flow cytometry using haplotype-specific antibodies. Chimerism may be determined by short tandem repeat polymorphisms. When there is a sex-mismatch between the donor and the recipient, assays based on determining the frequency of sex-chromosomes may be used. Testing may be altered by principal investigator or designee.
Number of donor human leukocyte antigen (HLA) detection | Up to day 56
  Donors with distinct HLA A or B antigens that can be detected by flow cytometry will be chosen. This will enable tracking of infused cells.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT04220684/ICF_000.pdf